CLINICAL TRIAL: NCT02118727
Title: Phase 2B Study of Memantine for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Therapy in Amyotrophic Lateral Sclerosis (TAME)
Acronym: TAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Richard J. Barohn, MD, Executive Vice Chancellor for Health Affairs, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAME-ALS FD003937-01; FDA (Other Grant/Funding Number: R01FD003937)
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Frontal Temporal Dementia
Keywords: ALS; FTD; Tau; pNF-H/C3
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Pick Disease of the Brain | interventions — Memantine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Memantine (Active Comparator): Up to 20 mg memantine taken by mouth twice a day for 36 weeks
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Up to 2 placebo tablets taken by mouth twice a day for 36 weeks
  Interventions: Drug: Placebo (for Memantine)

INTERVENTIONS:
Drug: Memantine — All randomized patients will be instructed to take one tablet once a day for the first two weeks from a blinded bottle that contains 10 mg tablets or matching placebo. At week three, patients will be instructed to take one tablet twice a day from the 10 mg bottle or matching placebo. At week five, patients will be instructed to take one tablet in the morning and two tablets in the evening from the 10 mg bottle or matching placebo. At week seven patients will be instructed to take two tablets twice a day from the 10 mg bottle or matching placebo.
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo (for Memantine) — All randomized patients will be instructed to take one tablet once a day for the first two weeks from a blinded bottle that contains 10 mg tablets or matching placebo. At week three, patients will be instructed to take one tablet twice a day from the 10 mg bottle or matching placebo. At week five, patients will be instructed to take one tablet in the morning and two tablets in the evening from the 10 mg bottle or matching placebo. At week seven patients will be instructed to take two tablets twice a day from the 10 mg bottle or matching placebo.
  Other Names: Sugar pill manufactured to mimic memantine 10 mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if memantine at up to 20 mg twice a day when used in conjunction with riluzole, can slow down the disease progression of patients with ALS including potentially improving their neuropsychiatric changes, as well as determine if serum biomarkers can be used both as a diagnostic and a prognostic marker in patients with ALS.

Funding Source: FDA - Orphan Products Development (OPD)

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disease that affects 30,000 Americans each year. Of these 30,000 Americans, it has been suggested that up to 50% will experience cognitive and behavioral changes in the form of frontotemporal dysfunction and up to 40% will meet criteria for frontotemporal dementia (FTD). Riluzole the only FDA approved agent for ALS extends a patient's lifespan by 2-3 months, and there are no proven therapies for the cognitive changes associated with ALS. More effective therapy for this universally fatal disease is desperately needed.

Results from an open label pilot trial of 20 patients treated with memantine at 10 mg twice a day suggested that treatment with the combination of memantine and riluzole slowed ALS disease progression. This trial also showed that levels of specific protein biomarkers in the cerebrospinal fluid (CSF) at baseline correlated with the rate of disease progression. A concurrent phase II study performed by Dr. Carvalho, found no effect with similar dosing; however, the study was limited in terms of power. Comments on previous failed drug trials in ALS have raised the concern that many ALS trials study a potential therapeutic agent at only a single dose and thus may miss the potential efficacy of non FDA approved doses; therefore, this proposed study will test a higher dose of memantine, 20 mg twice a day, in a double blind, placebo controlled, randomized trial of 90 patients with ALS to determine if a therapy of memantine, especially in combination with riluzole, can slow disease progression compared to treatment with riluzole alone or no treatment. Participants who experience treatment related adverse events may undergo dose reduction or discontinuation. The primary outcome measure will be the rate of disease progression as measured by the ALS Functional Rating Scale- Revised (ALSFRS-R). In addition the investigators will examine the cognitive deficits seen in ALS patients measured by the ALS Cognitive Behavioral Screen (ALS-CBS) and the Neuropsychiatric Inventory Questionnaire (NPI-Q). Finally the investigators will examine specific validated protein serum biomarkers to determine if there is a correlation between the levels of these biomarkers and the rate of disease progression. In particular the investigators will measure the ratio of phosphorylated heavy neurofilament to Complement 3 to see if this ratio is predictive of disease progression and if the levels change during therapy with memantine.

This project will offer unique insights into this untreatable disease. If this study confirms earlier results and suggests that memantine, when used in conjunction with riluzole, significantly slows down the progression of the disease, as well as ameliorates cognitive deficits in patients with fronto-temporal dysfunction, it will set the groundwork for conducting a larger phase III trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Male or Female
3. Clinically definite, probable, probable lab-supported, or possible ALS by El Escorial criteria
4. ALSFRS-R > 25
5. Must be willing to undergo longitudinal blood draws for biomarker analysis
6. Availability and willingness to complete the study
7. Capable of providing informed consent and complying with trial procedures
8. If patients are taking riluzole and/or Radicava, they must be a on a stable dose for at least thirty days prior to the baseline.

Exclusion Criteria:

1. Patients with forced vital capacity (FVC) ≤ 60%
2. History of liver disease
3. Severe renal failure
4. History of intolerance to memantine
5. Onset of weakness for greater than 3 years
6. Any other co-morbid condition which would make completion of the trial unlikely
7. If female, pregnant or breast-feeding; or, if of childbearing age, an unwillingness to use birth control.
8. Taking any investigational medications. If the patient was previously on investigational medications, a 30-day washout period is required before the baseline visit. Non-trial medications are not cause for exclusion.
9. Unwillingness to provide consent

Remote Inclusion Criteria:

1. Age 18-85
2. Male or Female
3. Clinically definite, probable, probable lab-supported, or possible ALS by El Escorial criteria
4. ALSFRS-R > 25
5. Must be willing to undergo longitudinal blood draws for biomarker analysis. This may be foregone during the screening visit
6. Availability and willingness to complete the study
7. Capable of providing informed consent and complying with trial procedures
8. If patients are taking riluzole and/or Radicava, they must be a on a stable dose for at least thirty days prior to the baseline
9. Documentation of not clinically significant liver enzymes within the previous 6 months

Remote Exclusion Criteria:

1. Patients with FVC ≤ 60%*
2. History of liver disease
3. Severe renal failure
4. History of intolerance to memantine
5. Onset of weakness for greater than 3 years
6. Any other co-morbid condition which would make completion of the trial unlikely
7. If female, pregnant or breast-feeding; or, if of childbearing age, an unwillingness to use birth control.
8. Taking any investigational medications. If the patient was previously on investigational medications, a 30-day washout period is required before the baseline visit. Non-trial medications are not cause for exclusion.
9. Unwillingness to provide consent

   * Since FVC cannot be captured during a remote screening visit, and acceptable FVC performed within the previous 90 days is acceptable. If an FVC is not available within the previous 90 days, the subject may be enrolled if the local site PI believes the subject has no significant shortness of breath or respiratory issues.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Barohn, MD, Principal Investigator — University of Missouri Health Care
Locations (13):
- United States (13):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - UC Irvine, Irvine, California
  - University of Florida, Jacksonville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas School of Medicine - Wichita, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Missouri, Columbia, Missouri
  - CoxHealth, Springfield, Missouri
  - Providence Health Sciences, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - Nerve & Muscle Center of Texas, Houston, Texas
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 58 | 31
Completed | 33 | 20
Not Completed | 25 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 58 | 31 | 89
Age, Continuous [Mean (Full Range); unit: years] | 62 [24 to 83] | 63 [38 to 81] | 63 [24 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 10 | 37
  Male | 31 | 21 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 53 | 30 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 58 | 31 | 89
ALSFRS-R [Mean (Standard Deviation); unit: units on a scale] — The Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) is a 12 question rating scale used to determine each participant's assessment of their capability and independence in daily activities. Possible values are from 0 to 48; higher score means better outcome.
  units on a scale | 36.33 (5.50) | 38.1 (5.37) | 36.94 (5.49)
Forced vital capacity (FVC) [Mean (Standard Deviation); unit: % of the predicted value] — Forced vital capacity % of the predicted value Population: Baseline FVC values were collected for 44/58 participants randomized to memantine and 27/31 participants randomized to placebo.
  % of the predicted value
    number analyzed (Participants) | 44 | 27 | 71
    (all) | 86.62 (15.51) | 82.02 (15.15) | 83.05 (18.82)
Symptom Duration [Mean (Standard Deviation); unit: Months] | 11.31 (5.44) | 11.61 (6.44) | 11.42 (5.77)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Comparison for Efficacy Will be Based on a Linear Mixed Effects (LME) Model Fit to the ALSFRS-R Data for the Patients Followed Over 36 Weeks.
Description: The primary outcome measure will be disease progression as measured by the Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) during the 36 weeks of therapy. The patient's rate of progression on active therapy during the 36 week treatment arm will be compared to the rate of progression of the placebo arm. The ALSFRS-R is a 12 question rating scale used to determine each participant's assessment of their capability and independence in daily activities. Possible values are from 0 to 48; higher score means better outcome.
Time Frame: During 36 weeks of therapy
Population: Includes the 54/58 participants randomized to memantine and 29/31 participants randomized to placebo with more than one ALSFRS-R value.
Measure: Mean (Standard Error); unit: score on a scale/week
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 54 | 29
score on a scale/week | -0.290 (0.39) | -0.281 (0.32)

2. Other Pre Specified Outcome: Measuring the Levels of Tau, Phosphorylated Neurofilament Heavy Chain (pNFH) and the pNFH/C3 Ratio in Blood
Description: Preliminary data have demonstrated that there are elevated levels of Tau and pNF-H in the blood of patients with ALS as compared to healthy controls suggesting that these proteins could also be used for measuring a patient's disease progression.
Time Frame: 36 weeks of treatment
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Slowing of Behavioral Decline in Those With FTD Characteristics Based on the NPI-Q and the ALS-Cognitive Behavioral Screen (CBS)™
Description: The ALS Cognitive Behavioral Screen (ALS-CBS™) and the Neuropsychiatric Inventory Questionnaire (NPI-Q), are two neuropsychological batteries that are validated measurements of frontotemporal dementia (FTD). The ALS-CBS questionnaire rates changes perceived in the patient by the caregiver. Possible values for the Cognitive score are from 0-20, and for the Behavior score are from 0-45. A higher score means better outcome. The NPI-Q provides an informant-based assessment of neuropsychiatric symptoms and associated caregiver distress for evaluating psychopathology in dementia. Possible values for the 12 item Total NPI score are from 0-36, and for the 12 item Total Distress score are from 0-30. A lower score means a better outcome
Time Frame: 36 weeks of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 40 weeks
Description: Adverse Events - Clinical abnormalities that begin or worsen and are not thought to be directly related to the expected course of ALS itself, whether or not the abnormality is believed by the investigator to be related to the study medication.
  Serious Adverse Events - Life threatening, fatal, result in hospitalization or prolong hospitalization, permanent disability, congenital anomaly, cancer, or overdose, or are any event that the investigator believes is very unusual or potentially serious.
Arm/Group | Memantine | Placebo
All-Cause Mortality (participants affected / at risk) | 3/58 | 3/31
Serious Adverse Events (participants affected / at risk) | 8/58 | 3/31
Other Adverse Events (participants affected / at risk) | 46/58 | 19/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=58) | Placebo (N=31)
Lung infection (Infections and infestations) | 3 (3) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=58) | Placebo (N=31)
Confusion (Psychiatric disorders) | 10 (10) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 15 (18) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 15 (28) | 5 (8)
Fatigue (General disorders) | 7 (7) | 0 (0)
Flu like symptoms (General disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3)
Muscular weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Ataxia (Nervous system disorders) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Pain (General disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT02118727/Prot_SAP_000.pdf